CLINICAL TRIAL: NCT03197051
Title: Impact of Perioperative Shedding of the Endothelial Glycocalyx on the Incidence of Postoperative Acute Kidney Injury in Patients Undergoing Valvular Heart Surgery.
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2017-0340
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Valvular Heart Disease
Keywords: Endothelial glycocalyx; Acute kidney injury; Valvular heart disease
MeSH Terms: conditions — Heart Valve Diseases; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Q1: Measure the Concentration of Syndecan-1, Heparan sulfate before anesthetic induction and immediately after weaning from cardiopulmonary bypass. Categorize the patients by serum syndecan-1 concentration(off-CPB) quartile. Q1 means a group of lowest 25% of serum syndecan-1 concentration.
- Q2: Q2 means a group of lower 25~50% of serum syndecan-1 concentration.
- Q3: Q3 means a group of higher 50~75% of serum syndecan-1 concentration.
- Q4: Q4 means a group of highest 75~100% of serum syndecan-1 concentration.

SUMMARY:
Endothelial glycocalyx, the luminal structure of healthy vasculature, plays critical roles in regulation of inflammatory responses, vascular permeability, blood coagulation. It can be easily damaged by ischemia/reperfusion, hypoxemia, oxidative stress, endotoxin. Accordingly, the relationship between the shedding of endothelial glycocalyx and the prognosis of diseases such as diabetes mellitus, atherosclerosis, malignancy has been researched.

In cases of cardiac surgery, patients cannot help but be exposed to ischemia/reperfusion, oxidative stress which can damage endothelial glycocalyx. In this research, the investigators would like to discover the impact of perioperative shedding of the endothelial glycocalyx on the incidence of postoperative acute kidney injury in patients undergoing valvular heart surgery.

DETAILED DESCRIPTION:
Syndecan-1, Heparan sulfate serve as biomarkers of glycocalyx degradation. Both biomarkers will be measured 2 times, before the anesthetic induction, and immediately after weaning from cardiopulmonary bypass, during the valvular heart surgery.

Postoperative acute kidney injury up to postoperative 48 hours, Composite morbidity and mortality up to postoperative 30 days will be checked.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing valvular heart surgery (>20 years old)

Exclusion Criteria:

* Emergency operation
* Aorta surgery (Graft replacement of Total arch or Descending thoracic aorta)
* Minimal invasive surgery
* Chronic kidney disease (eGFR<30mL/min/1.73m2) / Dialysis history
* Infective endocarditis
* Malignancy
* Patients who cannot give Informed consent (e.g. Illiterate, Foreigners)
* Patients who are already enrolled to another study than can affect the results

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing valvular heart surgery (>20 years old)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2017-06-25 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury | Up to Postoperative 48 hours
  Acute kidney injury is classified under KDIGO guideline.
  Stage I
  * Serum creatinine (Scr) : 1.5 to 1.9 times baseline or ≥26μmol/L (≥3.0mg/dL) increase
  * Urine output : <0.5mL/kg/kr for 6~12hrs
  Stage II
  * Serum creatinine (Scr) : 2.0 to 2.9 times baseline
  * Urine output : <0.5mL/kg/hr for ≥12hrs
  Stage III
  * Serum creatinine (Scr) : 3.0 times baseline or ≥354μmol/L (≥4.0mg/dL) increase or Initiation for RRT
  * Urine output : <0.3mL/kg/hr for ≥24hrs or Anuria for ≥12hrs

SECONDARY OUTCOMES:
Composite morbidity and mortality (by STS Major morbidity endpoint) | Up to postoperative 30 days
  STS Major morbidity endpoint
  * Mortality for postoperative 30 days irrelevant to causes
  * Permanent stroke
  * Wound infection
  * Prolonged ventilation greater than 48 hours
  * Cardiac surgery reoperation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No